CLINICAL TRIAL: NCT05490537
Title: Clinical Evaluation of the Cutaneous Acceptability, Comedogenic Potential and Efficacy of Two Cosmetic Products Used in Synergy
Brief Title: Cutaneous Acceptability, Comedogenic Potential and Efficacy of Two Cosmetic Products Used in Synergy
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: LRP19013-EFFACLAR GEL AND DUO+
Record Dates: First submitted 2022-08-02; First posted 2022-08-05 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Acne
Keywords: acne; comedogenic potential; GEA
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The open, intra-individual study aims to assess the cutaneous acceptability, comedogenic potential and efficacy of a cleansing gel and a cream used in synergy to relieve patients presenting with acne grade 2 and 3. Each subject is her/his own control.

DETAILED DESCRIPTION:
The evaluation of Effaclar gel and Effaclar Duo+ used in synergy in acneic patients has been conducted under dermatological control by Dermscan that is certified by the International Standards Organization (ISO) 9001-2015.

Each study report is subjected to a quality inspection by a member of Dermscan. A certificate of quality inspection signed by the proofreader (not involved in the study) who checked the report is enclosed in each study. The inspection of the study report allows to confirm that the results reflect exactly the study raw data and that the study fulfills any standard and regulatory requirements.

With regard to the statistical analysis, and in particular the descriptive analysis, each quantitative criterion and scores will be summarized using the following standard statistics

* number of valid values
* number of missing values,
* means,
* standard deviations,
* standard errors of the mean,
* medians,
* minimum values and
* maximum values for each time point by product. The qualitative data will be summarized in frequency (N) and percentage (%).

With regard to the statistical analysis, and in particular the inferential analysis, for each quantitative assessed criterion, a mixed ANOVA model for repeated measurements (fixed factors included: product with 2 levels and time with 3 levels) will be fitted to raw data.

To take into account the correlation between data obtained from a same subject, an unstructured variance -covariance matrix (UN@UN) will be set.

The specific contrasts of interest on adjusted means (LS-Means) will be built:

* to assess the change on (Di) from baseline (D0) for each product
* to test whether products differ significantly in terms of change from baseline (Di-D0).

The participants have the right to exit from the study at any time and for any motive in compliance with the Helsinki Declaration (1964) and its successive updates. The investigator can also interrupt the person's participation in the study prematurely in the case of a disease occurrence, a pregnancy or the occurrence of an adverse reaction.

Every premature exit must be classified under one of the following headings:

* presence of a non-inclusion criteria;
* Undesirable Effect / Adverse Event occurrence;
* Serious Adverse Event / Serious Adverse Effect occurrence;
* withdrawal of consent;
* lost to follow-up;
* appearance of non-inclusion criteria;
* non-adherence to the protocol;
* other reason. All the adverse events and serious adverse events are reported in the case report form and the study report.

  70 persons have been pre-included in order to include 46 participants and to obtain results on 42 (±10%) participants minimum in each centre (2 centers in total).

The personnel in charge of the study collects data into individual case report forms in electronic or paper format and/or directly from measurement software. When information is collected in paper format, the simple/double data entry is then done from these supports by the designed operator(s), without any interpretation, in specific EXCEL databases. The Project Manager or assistant checks the double data entry by comparing both databases.

Then the coherence of the whole data set is checked as well as formulas used in the EXCEL tables (calculation formulas, selected data…).

When all the controls are done, the database is locked.

ELIGIBILITY:
Inclusion Criteria:

* phototype I to VI according to the following distribution:

  * 7 female subjects of <18 years old and phototype I or II, 7 male subjects of <18 years old and phototype I or II, 7 female subjects of >18 years old and phototype I or II, 7 male subjects of >18 years old and phototype I or II,
  * 7 female subjects of <18 years old and phototype III or IV, 7 male subjects of <18 years old and phototype III or IV, 7 female subjects of >18 years old and phototype III or IV, 7 male subjects of >18 years old and phototype III or IV,
  * 7 female subjects of <18 years old and phototype V or VI, 7 male subjects of <18 years old and phototype V or VI, 7 female subjects of >18 years old and phototype V or VI, 7 male subjects of >18 years old and phototype V or VI
* Caucasian (in Dermscan in Poland) and Negroid (in Insight Research in Mauritius)
* participants with GEA (Global Evaluation Acne) 2 or 3 at inclusion
* Participants with at least 15 retentional and 7 inflammatory lesions on the face at the inclusion.

Exclusion Criteria:

* cutaneous pathology on the studied zone other than acne (eczema, ...)
* topical acne treatment since less than one month
* participant manipulating her/ his acne lesions
* excessive exposure to sunlight or UV-rays within the previous month
* use of topical or systemic treatment during the previous weeks liable to interfere with the assessment of the acceptability and efficacy of the studied products (according to the investigator's appreciation)

Max Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: participants with acne grade 2 and 3 meeting the inclusion and exclusion criteria and agreeing to the study contraints
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
change in cutaneous acceptability by the dermatologist with a 5-point scale | from baseline to Day56
  assessment of the acceptability of the parameters erythema, edema, dryness, desquamation, roughness on a 5-point scale (none, very mild, mild, moderate, severe)
change in cutaneous acceptability by the participant with a 5-point scale | from baseline to Day56
  assessment of the acceptability of the parameters tightness, stinging, itching, warm/burning sensation on a 5-point scale (none, very mild, mild, moderate, severe)
change in comedogenic potential | from baseline to Day56
  The variations (Day28-Day0, Day56-Day0) in the number of lesions are calculated for each kind of lesions. Descriptive statistics are done in order to determine the variation significance.
  * a non-comedogenic product does not induce any significant increase in the number of retentional lesions.
  * a non-acnegenic product does not induce any significant increase in the number of inflammatory lesions.
change in Global Evaluation Acne (GEA) score | from baseline to Day56
  The dermatologist realizes clinical score of the product's anti-acne efficacy using the Investigator Global Acne Severity Score with a 6-point scale: from 0 Clear. No lesions. to 5. Very severe

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Bednarczyk, Study Director — Eurofins
Locations (2):
- Insight Research, Quatre Bornes, Mauritius
- Dermscan Poland Sp. z o. o., Gdansk, Poland